CLINICAL TRIAL: NCT00269776
Title: Screening, Efficacy, and Safety Study Evaluating OROS (Methylphenidate HCl), Ritalin and Placebo in Children With ADHD
Brief Title: An Effectiveness and Safety Study Evaluating OROS Methylphenidate Hydrochloride (HCl), Ritalin (Methylphenidate HCl) and Placebo in Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: Director, Clinical Research - CNS, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR005989; CONCERTAATT3019; C-98-003-02
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; OROS; children; methylphenidate; Ritalin
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 001 (Experimental): OROS (methylphenidate HCl) Treatment A: 1 2 or 3 OROS methylphenidate 18-mg tablets + 0 1 or 2 OROS placebo tablets (3 tablets in total) once daily + 1 placebo capsule 3x/day for 7 days. Each patient will be randomized to 1 of 9 treatment sequences each consisting of 3 7-day treatment periods of Treatment A B and C.
  Interventions: Drug: OROS (methylphenidate HCl)
- 002 (Experimental): Ritalin (methylphenidate) Treatment B: 5 10 or 15-mg tablets (encapsulated/single capsule) 3 times a day + 3 OROS placebo tablets once daily for 7 days. Each patient will be randomized to 1 of 9 treatment sequences each consisting of 3 7-day treatment periods of Treatment A B and C.
  Interventions: Drug: Ritalin (methylphenidate)
- 003 (Experimental): Placebo Treatment C: Three OROS placebo tablets once daily + 1 placebo capsule 3x times/day for 7 days. Each patient will be randomized to 1 of 9 treatment sequences each consisting of 3 7-day treatment periods of Treatment A B and C.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Treatment C: Three OROS placebo tablets once daily + 1 placebo capsule 3x times/day for 7 days. Each patient will be randomized to 1 of 9 treatment sequences each consisting of 3 7-day treatment periods of Treatment A, B, and C.
  Arms: 003
Drug: OROS (methylphenidate HCl) — Treatment A: 1, 2, or 3 OROS methylphenidate 18-mg tablets + 0, 1, or 2 OROS placebo tablets (3 tablets in total) once daily + 1 placebo capsule 3x/day for 7 days. Each patient will be randomized to 1 of 9 treatment sequences each consisting of 3 7-day treatment periods of Treatment A, B, and C.
  Arms: 001
Drug: Ritalin (methylphenidate) — Treatment B: 5, 10, or 15-mg tablets (encapsulated/single capsule) 3 times a day + 3 OROS placebo tablets once daily for 7 days. Each patient will be randomized to 1 of 9 treatment sequences each consisting of 3 7-day treatment periods of Treatment A, B, and C.
  Arms: 002

SUMMARY:
The purpose of this study is to provide data on the effectiveness of the OROS Methylphenidate Hydrochloride (HCl) formulation compared to placebo and standard immediate-release Ritalin with respect to improving attention and behavior, and decreasing hyperactivity in children with Attention Deficit Hyperactivity Disorder (ADHD). Both OROS Methylphenidate HCl and Ritalin contain the central nervous system stimulant, methylphenidate HCl. The safety associated with the two methylphenidate formulations will also be compared with placebo.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) represents the most common neurobehavioral disorder in children, affecting 3% to 5% of the school-age population. Behavioral pediatricians, child psychiatrists, and child neurologists indicate that referrals for ADHD may constitute up to 50% of their practices. This is a double-blind, double-dummy, randomized, placebo-controlled, active-controlled, 3-treatment, 3-period crossover trial to compare the safety and effectiveness (onset of effect, time to loss of effect and overall efficacy) of OROS Methylphenidate Hydrochloride (HCl), with standard immediate-release Ritalin and placebo. During this study, patients receive each of the three treatments (OROS Methylphenidate HCl 18, 36 or 54 milligrams per day, Ritalin 5, 10 or 15 milligrams three times per day, or placebo) for 7 days, and are assigned to one of three dosage levels depending upon their prestudy methylphenidate dose and regimen. The total study participation for each patient will be 21 days. Since ADHD is manifested in a variety of settings and can affect attention and behavior, this study assesses efficacy in home, community school, and laboratory school settings using numerous assessments designed to evaluate various aspects of the disorder. These assessments are completed by a variety of raters, including the parents/caregivers, community school teachers, and laboratory school teachers. The primary measure of effectiveness is the community school teacher's rating on the IOWA Conners Inattention/Overactivity subscale. Additional measures of effectiveness include the IOWA Conners (Inattention/Overactivity and Oppositional/Defiance subscale) ratings, SKAMP attention and deportment ratings, peer interaction and other behavioral ratings, global assessments, SNAP-IV ratings, activity levels during structured activities, accuracy and productivity of independent assigned academic seatwork, and a home situation questionnaire. Safety evaluations include the incidence of adverse events, physical examinations, clinical laboratory tests, vital signs, sleep quality, actigraphy (sleep latency, duration, and arousals), appetite, and the presence/severity of tics (hard-to-control, repeated twitching of any parts of the body or hard-to-control repeating of sounds or words). Patients will be given oral doses of: OROS (methylphenidate HCl) 1, 2, or 3 of the 18-milligram tablets once daily, or Ritalin 5, 10, or 15 mg (encapsulated/single capsule) three times a day, or placebo. There are three treatment groups, each group dosing for 7 days for a total of 21 days on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients having a diagnosis of one of the three subtypes of Attention Deficit Hyperactivity Disorder (ADHD) verified by both a parent/child interview and a teacher assessment using SNAP-IV questionnaires
* taking or have taken in the past 5 - 20 mg of immediate-release methylphenidate (Ritalin) at least twice a day, 20 - 60 mg of sustained-release methylphenidate (Ritalin-SR) per day, or a combination of immediate-release and sustained-release methylphenidate up to a daily dose not exceeding 60 mg
* having used methylphenidate for at least 3 months at some time in the past without any significant adverse experiences, considered to be positive responders to methylphenidate therapy, and agreeing to take to take only the supplied study drug as treatment for ADHD during the three-week treatment phase of the study
* able to comply with the study visit schedule and whose parent(s) and teacher are willing and able to complete the protocol-specified assessments
* agreeing not to ingest any caffeine containing beverages (e.g., coffee or soda) or foods (e.g., chocolate) on days 7, 14, and 21 of the study.

Exclusion Criteria:

* Patients having clinically significant gastrointestinal problems, including narrowing of the gastrointestinal tract
* having glaucoma, an ongoing seizure disorder, a psychotic disorder, or have a diagnosis of Tourette's syndrome
* whose primary treatment focus is oppositional-defiant disorder, conduct disorder, or tics, or whose primary treatment focus is psychiatric conditions such as depressive disorders, bipolar disorders, or other mood disorders
* having a mean of two blood pressure measurements (systolic or diastolic) equal to or greater than the 95th percentile for age, sex, and height at screening
* if female, have begun menstruation.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1998-11; Study Completion 1999-01 (Actual)

PRIMARY OUTCOMES:
IOWA Conners Inattention/Overactivity subscale ratings by the Community School Teacher | Up to Day 6 of each treatment period for a total of approximatly 18 days

SECONDARY OUTCOMES:
SKAMP attention and deportment ratings | Up to Day 7 of each of 3 treatment periods for a total of approximately 21 days
Peer interaction ratings | Up to Day 7 of each of 3 treatment periods for a total of approximately 21 days
Laboratory School Teacher Global Assessments | Up to Day 7 of each of 3 treatment periods for a total of approximately 21 days
SNAP-IV ratings | Up to Day 7 of each of 3 treatment periods for a total of approximately 21 days
Incidence of adverse events | Up to Day 7 of each of 3 treatment periods for a total of approximately 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA

REFERENCES:
- [Result] Swanson J, Gupta S, Lam A, Shoulson I, Lerner M, Modi N, Lindemulder E, Wigal S. Development of a new once-a-day formulation of methylphenidate for the treatment of attention-deficit/hyperactivity disorder: proof-of-concept and proof-of-product studies. Arch Gen Psychiatry. 2003 Feb;60(2):204-11. doi: 10.1001/archpsyc.60.2.204. PMID 12578439